CLINICAL TRIAL: NCT05946733
Title: Comparison Between The Analgesic Effect of Oblique Subcostal and Lateral Approach of Ultrasound-Guided Transverse Abdominis Blocks for Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Two Approaches of Transversus Abdominis Block (TAP ) in Laparoscopic Cholecystectomy
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, Lecturer of Anesthesiology, Intensive Care and Pain Management Faculty of Medicine - Menoufia University, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11/2022ANET10-26
Record Dates: First submitted 2023-06-17; First posted 2023-07-14 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into three equal groups using SPSS. Group A: will receive bilateral oblique subcostal TAP block Group B: will receive bilateral lateral TAP block. GroupC:will receive postoperative morphine by patient-controlled analgesia (PCA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): subcostal TAP block
  Interventions: Procedure: Group A
- Group B (Experimental): lateral TAP block.
  Interventions: Procedure: Group B
- GroupC (Other): will receive postoperative morphine by patient-controlled analgesia (PCA).
  Interventions: Other: Group C

INTERVENTIONS:
Procedure: Group A — After induction of general anesthesia, oblique subcostal TAP blocks will be done(14) under the guidance of Sonosite ,superficial probe ,14-15 MHz ultrasound transducer
  Arms: Group A
Procedure: Group B — After induction of general anesthesia, bilateral lateral TAP block will be performed (15) under ultrasonographic guidance with transportable ultrasound device ( Sonosite ,superficial probe ,14-15 MHz)
  Arms: Group B
Other: Group C — the analgesia will be maintained using a morphine patient-controlled analgesia (PCA) device set to give 1.5 mg bolus administration of morphine without a basic rate and 15 min lock-out time. The total amount of morphine administration will be recorded for the subsequent 24 h
  Arms: GroupC

SUMMARY:
the investigators will compare the effect of pre-operative oblique subcostal TAP and lateral TAP blocks on the total perioperative opioids consumption for patients undergoing elective laparoscopic cholecystectomy

DETAILED DESCRIPTION:
General anesthesia induction will be achieved using a sleeping dose of fentanyl 1µg/kg intravascular(IV), propofol 2mg/kg (IV), and atracurium 0.5mg/kg (IV) to facilitate tracheal intubation. General anesthesia will be maintained with lungs ventilation by pressure controlled mode with isoflurane

During anesthesia maintenance Intraoperatively, if blood pressure BP or heart rate (HR) increase more than 20% from baseline, intravenous morphine (3- 5mg) will be given to stabilize the patients' haemodynamics. Fifteen minutes before the end of surgery all patients will receive 1g intravenous paracetamol and 4 grams ondansetron.

Patients will be randomly divided into three equal groups:

Group A: will receive bilateral oblique subcostal TAP block Group B: will receive bilateral lateral TAP block. Group C :will receive postoperative morphine by patient-controlled analgesia (PCA).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be older than 21 years old with American society of anaesthesia physical status I& II scheduled for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* - Uncooperative.
* Patients who have allergy to any of the study drugs.
* Patients who are on opioids.
* Known abuse of alcohol or medication.
* Local infection at the site of injection or systemic infection.
* Pregnancy.
* Patients with coagulation disorders or on anticoagulation therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-26 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 48 hours
  milligrams

SECONDARY OUTCOMES:
patient satisfaction | 48 hours
  visual analogue scale ((a scale from 0 to 10 where 0 is interpreted as no pain, 1-4 mild pain, 5-6 moderate pain, 7-10 severe pain)
anesthesia recovery time | 1hour
  minutes
total perioperative analgesics requirements | 24 hours
  milligrams
Post-operative anaesthetic care unit (PACU) stay | 2 hours
  minutes

CONTACTS AND LOCATIONS:
Overall Officials: AMAL G SAFAN, MD, Study Director — Menoufia University
Locations (1):
- Menoufia University, Cairo, Shibin Elkom, Egypt